CLINICAL TRIAL: NCT05895201
Title: Phase I/II Trial of High-Dose Post-Transplant Cyclophosphamide, Bortezomib, and Sitagliptin for the Prevention of Graft-versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: High-Dose Post-Transplant Cyclophosphamide, Bortezomib, and Sitagliptin for the Prevention of GVHD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI has left IU with no plan to initiate study at IU
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0778
Record Dates: First submitted 2023-05-19; First posted 2023-06-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-10

CONDITIONS: Bone Marrow Transplant Complications; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia, Adult; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
Keywords: Allogenic peripheral blood stem cell grafts; Phase I; Phase II
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Sitagliptin Phosphate; Bortezomib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sitagliptin + Bortezomib + Cyclophosphamide (Experimental)
  Interventions: Drug: Sitagliptin; Drug: Bortezomib; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Sitagliptin — 600 or 400 (or MTD) mg PO every 12 hours on days -1 to +14 depending on dose level assignment.
Drug: Bortezomib — 1.3 or 1.0 mg/m2 (or MTD) IV push 6 hours after graft infusion completion (day 0), and 72 hours thereafter depending on dose level assignment.
Drug: Cyclophosphamide — 50 mg/kg IV over 1 hour on days +3 and +4

SUMMARY:
This is an open label Phase I-II study to determine the safe doses of bortezomib, sitagliptin, and PTCy (Phase I) with expansion into a phase II trial to determine efficacy in improving survival.

DETAILED DESCRIPTION:
Determine the safe doses of bortezomib, sitagliptin, and PTCy for use in expansion into a phase II trial. This is effectively the maximum tolerated dose of the drugs tested in a 3+3 design in a limited phase I portion. Phase I requires a maximum of 18 patients.

Determine the efficacy of sitagliptin, bortezomib, and PTCy in improving the survival free of grade II-IV acute GVHD at day +100 from an expected 65% to 80% or more. This portion uses a Simon minimax two-stage design, testing the null hypothesis H0: p0 < 0.65 versus the alternative hypothesis H1: p1 ≥ 0.8, where p is the probability of being alive and without grade II-IV acute GVHD at day 100 after transplantation. Using a minimax optimal stage design with a one-sided type I error set to 0.05, and a type II error rate set to 0.2 (power 80%). In the first stage, 31 evaluable patients will be entered. If 20 or fewer are alive without acute grade II-IV GVHD (i.e., 11 or more develop acute grade II-IV GvHD) by day +100, the study will be stopped in favor of the null hypothesis. On the other hand, if more than 20 are alive without grade II-IV acute GVHD by day +100, and additional 24 patients will be enrolled for a total of 55 evaluable patients. In the final analysis, if more than 41 remain alive free of grade II-IV acute GVHD (i.e., only 14 or less have developed acute grade II-IV acute GVHD by day +100), the null hypothesis will be rejected, and will conclude that the combination used for prevention of moderate to severe GVHD is worthy of further study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any of the following hematologic malignancies:

   * Acute myeloid leukemia (AML) in first remission (CR1) if they have with intermediate or high-risk cytogenetic and/or molecular features, or patients in second or subsequent complete remission (CR2, CR3, etc.). Complete remission is defined as presence of <5% blasts in the bone marrow Version 09/30/2022 25 with no morphological evidence of leukemia. Patients in CR with incomplete count recovery may be included.
   * Acute lymphoblastic leukemia (ALL) with any of the following in CR1 or subsequent complete remission (CR2, CR3, etc.). Complete remission is defined as presence of <5% blasts in the bone marrow with no morphological evidence of leukemia. Patients in CR with incomplete count recovery may be included.
   * Myelodysplastic disorder (MDS) with a revised International Prognostic System Score (IPSS-R)104 of greater than 3 at diagnosis. Patients must have <10% blasts in the bone marrow documented within 30 days of transplant.*
   * Therapy-related myelodysplastic disorder (t-MDS). Patients must have <10% blasts in the bone marrow documented within 30 days of transplant.*
   * Chronic myelomonocytic leukemia (CMML) type 1 or 2. Patients must have <10% blasts in the bone marrow documented within 30 days of transplant.* *Patients with MDS, t-MDS, and CMML will be included only in the phase I portion of the study.
2. Patient age ≥ 18 years
3. Karnofsky Performance status ≥ 70%
4. Patients must also be suitable to receive a reduced-intensity (RIC) conditioning regimen at the discretion of the treating physician. While there are not universally accepted or validated cut-off criteria of age, performance status, or hematopoietic cell transplantation-comorbidity index (HCT-CI) for suitability for RIC, RIC transplants should be considered for patients 60 years and older, and for patients <60 years who are "less fit", e.g., KPS <90% and/or HCT-CI ≥ 3 due to lower non-relapse mortality associated with RIC.
5. Patients receiving allogeneic peripheral blood stem cell (PBSC) grafts from HLA-matched (5/6 and 6/6 matches) siblings or matched unrelated donors (7/8 or 8/8 matches at HLA-A, B, C, DRB1 by high resolution typing) are included. All grafts will be unmanipulated (i.e., no T cell depleted or CD34 selected grafts). In addition, donors should meet institutional criteria for donation of PBSC, as well as the screening and eligibility criteria of the National Marrow Donor Program (NMDP) for unrelated donors, and the requirements of the United States Food and Drug Administration for Human Cell, Tissue, or Cellular or Tissue-based Products (HCT/P) (21 CFR Part 1271).
6. Required baseline laboratory values within 16 days prior to admission:

   * Estimated creatinine clearance >60 ml/min/1.72 m2
   * Serum total bilirubin ≤ 2 x upper limit of normal value (except for Gilbert's disease)
   * AST and ALT ≤ 3 x upper limit of normal value
   * Alkaline phosphatase (ALP) ≤ 250 IU/l
7. Required baseline values within 60 days prior to admission:

   * Left ventricular ejection fraction (LVEF) >40% Version 09/30/2022 26
   * Adjusted carbon monoxide diffusing capacity (DLCO) >50%
8. No evidence of HIV infection (Patients with immune dysfunction are at a significantly higher risk of infection from intensive immunosuppressive therapies.)
9. Non-pregnant and non-nursing
10. Signed written informed consent
11. Patients must otherwise fulfill institutional criteria for eligibility to undergo reduced-intensity allogeneic stem cell transplantation.

Exclusion Criteria:

1. Pregnant or nursing females or women of reproductive capability who are unwilling to completely abstain from heterosexual sex or practice 2 effective methods of contraception from start of conditioning through a minimum of 90 days after the last dose of study drug.
2. Male subjects who refuse to practice effective barrier contraception from the start of conditioning through a minimum of 90 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
3. Inability to provide informed consent.
4. Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
5. Patients with active central nervous system leukemia
6. Prior allogeneic HSCT or an autologous hematopoietic stem cell transplant in past 12 months
7. Patients with diabetes mellitus requiring insulin secretagogues and/or insulin at time of enrollment.
8. Patients with a history of pancreatitis
9. Patients with symptomatic cholelithiasis
10. Known hypersensitivity to any of the components of the investigational treatment regimen.
11. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
12. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma, an in-situ malignancy, or low-risk prostate cancer after curative therapy.
13. Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
14. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | in the first 30 days post-transplant
proportion of patients developing grades 3-4 non-hematological toxicity defining DLT assessed by CTCAE version 5.0 | in the first 30 days post-transplant
Proportion of patients alive and free of grade II-IV acute GVHD (graft-versus-host disease) | Baseline to day +100
Cumulative incidence of grade II-IV acute GVHD | through study completion (i.e. up to 5 years)

SECONDARY OUTCOMES:
Frequency of Non-Hematological toxicity as assessed by CTCAE version 5.0 | baseline to day +30
Cumulative incidences of all grades of acute GvHD | baseline to day +100
Chronic graft-versus-host disease | through study completion (i.e. up to 5 years)
Time to engraftment of neutrophils | the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (NEUTROPHILS + BANDS) is at least 0.5 x109/l.
Time to engraftment of platelets | the time to engraftment of platelets is defined as the time from day 0 to the first of seven consecutive days after transplantation during which the platelet count is at least 20 x109/l without transfusion support.
Cumulative Incidence engraftment of neutrophils and platelets | day 0 to the first of seven consecutive days after transplantation during which the platelet count is ≥ 20 x109/l and ANC is ≥ 0.5 x109/l without transfusion.
cumulative incidence of non-relapse mortality | through study completion (i.e. up to 5 years)
cumulative incidence of relapse | through study completion (i.e. up to 5 years)
Graft-versus-host free, and relapse-free survival (GRFS) | Baseline to day+365
chronic GvHD immunosuppression-free survival | Baseline through day+365
Grade III-IV acute GvHD-free survival | baseline through day +180
Progression-free Survival in all enrolled subjects | Baseline through day+365
Overall Survival in all enrolled subjects | Baseline through day+365

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States